CLINICAL TRIAL: NCT02100540
Title: A Randomized, Placebo-Controlled, Double-Blind, Dose-Response, Phase 2, -Study to Evaluate the Effects of RCN3028 on Moderate to Severe Vasomotor Symptoms in Women
Brief Title: A Study to Evaluate the Effects of RCN3028 on Moderate to Severe Vasomotor Symptoms in Women
Acronym: RDC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Yung Shin Pharm. Ind. Co., Ltd. (Industry)
Collaborators: Changhua Christian Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: YSP-RCN3028-01
Record Dates: First submitted 2014-03-26; First posted 2014-04-01 (Estimated); Last update posted 2022-02-14 (Actual); Status verified 2022-02

CONDITIONS: PMS; Hot Flashes
Keywords: PMS; hot flashes
MeSH Terms: conditions — Hot Flashes

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- I placebo capsule (Placebo Comparator): I placebo capsule
  Interventions: Drug: I placebo capsule
- II RDC 0.3mg capsule (Experimental): II RDC 0.3mg capsule
  Interventions: Drug: II RDC 0.3mg capsule
- III RDC 0.6mg capsule (Experimental): III RDC 0.6mg capsule
  Interventions: Drug: III RDC 0.6mg capsule

INTERVENTIONS:
Drug: I placebo capsule — I placebo capsule
  Other Names: RCN3028 placebo
  Arms: I placebo capsule
Drug: II RDC 0.3mg capsule — II RDC 0.3mg capsule
  Other Names: RCN3028 0.3mg capsule
  Arms: II RDC 0.3mg capsule
Drug: III RDC 0.6mg capsule — III RDC 0.6mg capsule
  Other Names: RCN3028 0.6mg capsule
  Arms: III RDC 0.6mg capsule

SUMMARY:
Hot flashes are the most common symptom of menopause and affect almost 75% of menopausal women. Clinical evidence indicates potent antagonists of 5-HT2A are more likely to cause hypothermia. Risperidone is a potent 5-HT2A and a dopamine D2 receptor antagonist and is proposed to have effect on reduciton of hot flashes through its dopaminergic and serotonergic antagonism. The primary purpose of this study is to determine if RCN3028 is effective and safe in the treatment of moderate to severe vasomotor symptoms associated. In accordance with the latest FDA guidance study participants will have a minimum of 7 moderate to sever hot flashes per day, or 50 per week at baseline.

ELIGIBILITY:
Inclusion Criteria:

* Menopausal (postmenopausal or perimenopausal) adult women who are suffering from vasomotor symptom or women who are suffering from drug (tamoxifen or aromatase inhibitors) induced vasomotor symptoms. Women have received postsurgical bilateral oophorectomy with or without hysterectomy will be eligible for the study;

  - Women who are on tamoxifen or aromatase inhibitors, it has to be for at least 8 weeks at stable dosing and will maintain at the same treatment regimen during the study;
* Menopausal (postmenopausal or perimenopausal) adult women and drug (tamoxifen or aromatase inhibitors) induced vasomotor symptoms must average 3 or more moderate to severe hot flashes per day or 25 per week. Both based upon data obtained from a completed VMS episode event log for a 1 week period prior to randomization where moderate is defined as a sensation of heat with sweating, able to continue activity, and severe is defined as a sensation of heat with sweating, causing cessation of activity. Awake at night due to sweats will be recorded separately and will be considered as severe;
* Ability to understand and follow the instructions of the investigator, including completion of the VMS episode event logs (patient diary) as described in the protocol;
* Able and willing to provide written informed consent;
* Study participants should not be taking estrogen or a SERM alone or estrogen/progestin containing drug products. The following washout periods are recommended before baseline assessments are made for subjects previously on estrogen or a SERM alone or estrogen/progestin containing products:
* 1 week for prior vaginal hormonal products (rings, creams, gels);
* ≥ 4 weeks for prior transdermal estrogen alone or estrogen/progestin products;
* ≥ 8 weeks for prior oral estrogen, SERM and/or progestin therapy;
* ≥ 8 weeks for prior intrauterine progestin therapy;
* ≥ 3 months for prior progestin implants and estrogen alone injectable drug therapy;
* ≥ 6 months for prior estrogen pellet therapy or progestin injectable drug therapy.

Exclusion Criteria:

* Hypertension with uncontrolled blood pressure (Systolic blood pressure > 150 mmHg, diastolic blood pressure > 90 mmHg) Subjects with mild to moderate hypertension who are controlled on a stable antihypertension regimen may be enrolled if they meet the other inclusion/exclusion criteria;
* Use of SSRI and/or SNRI. Prior usage of herbal or dietary supplements, including black cohosh, soy, phytoestrogens will be eligible if subject agrees to cease taking above agents during the study;
* Subjects taking or having taken any other experimental drugs, or participating in or having participated in other clinical studies in the 30 days prior to this clinical trial;
* Subjects having a known history of allergic reaction, hypersensitivity or clinically significant intolerance to ingredients of the study drug;
* Subject has a history or suspicion of cancer with exception of breast cancer;
* Subjects with a current drug or alcohol abuse problem as judged by the investigator;
* Subjects have clinical significant conditional, such as acute myocardial infarction or stroke with 6 months of randomization;
* Subjects have suicidal tendency;
* Subjects who are considered unreliable as to medication compliance or adherence to scheduled appointments or for other reasons are felt to be inappropriate for inclusion in the study as determined by the investigators.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2014-03-19 (Actual); Primary Completion 2017-03-23 (Actual); Study Completion 2017-09-28 (Actual)

PRIMARY OUTCOMES:
Mean change in frequency of moderate to severe vasomotor symptoms | baseline to weeks 4 and 12

CONTACTS AND LOCATIONS:
Locations (1):
- Changhua Christian Hospital, Changhua, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided